CLINICAL TRIAL: NCT04081896
Title: Evaluation of the Effects of Exercise-based Rehabilitation in Individuals with Spine Pain
Brief Title: Evaluation of the Effects of a Rehabilitation Program in Individuals with Spine Pain
Status: Recruiting | Type: Observational
Sponsor: SpineZone Medical Fitness, Inc (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kamshad Raiszadeh, MD, Principal Investigator, SpineZone Medical Fitness, Inc
Other Study IDs: Spine Exercise
Record Dates: First submitted 2019-04-16; First posted 2019-09-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Neck Pain; Low Back Pain; Scoliosis; Thoracic Injuries
MeSH Terms: conditions — Neck Pain; Low Back Pain; Scoliosis; Thoracic Injuries | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- In Clinic Rehabilitation: Participants who are undergoing supervised exercise based rehabilitation in the SpineZone clinic
  Interventions: Other: Exercise
- Online Rehabilitation: Participants who will be undergoing online-based coaching and exercise as prescribed via telephone, online chat, or web-based interactions with SpineZone rehabilitation staff (physical therapists and physicians)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise prescribed to participants includes spine-specific strengthening exercises targeting core musculature (i.e. Multifidus, Erector Spinae, Transversus Abdominus, Obliques, and Rectus Abdominus). The in-clinic exercise program recommends a minimum of 20 visits at 2 visits/week, with a goal of 24 total visits over a 12-week period. Exercise is progressed by 5-10% of their exercise load once they are able to do >20 repetitions. If they are able to reach >10 but <20 repetitions, exercise load remains the same. If they are unable to reach 10 repetitions, exercise load is decreased 5-10% at their next visit.
  The online exercise program includes non-machine based home exercises targeting the same muscles of interest, and are personalized to each participant based on their home resources and comfort level.
  Concurrent interventions may or may not include nutrition education, mindfulness, cognitive behavioral therapy.

SUMMARY:
SpineZone is an innovative physical therapy program with its focus on treatment of cervical, thoracic, and lumbar conditions through the use of a multi-disciplinary, technology enabled platform. Standard physical therapy modalities including psychologically informed physical therapy are employed in addition to online coaching with a fundamental tenant of core strengthening. Treatments are tracked and modified in a multi-disciplinary format taking all radiographic studies into direct consideration. The goal of this study is to utilize a registry of participants undergoing either in-clinic or online rehabilitation treatment for spine pain at the SpineZone clinical in order to understand the clinical outcomes and costs of different rehabilitation modalities in this patient population.

DETAILED DESCRIPTION:
The key objectives for this registry are to 1) identify magnitudes of clinical improvements with this specific specialized rehabilitation program in its various formats (in-clinic vs online), in individuals with or without spine pain for comparison to literature-based standard of care values for other conservative care protocols, 2) to identify average value of this treatment approach based on cost assessment, 3) to identify which patients (based on patient-specific predictors) are most likely to succeed with this specialized program and 4) to identify targets for improvement and optimization of patient care any necessary modifications to the industry's standard for care protocol. The goal of this project is to assess the impact of a standardized program based on core strengthening using technologic monitoring in a multidisciplinary format.

This registry of data will not contain individual identifiers.

The study population is comprised of skeletally mature patients, both male and female, from a wide variety of ethnicities representative of the typical population presenting with spinal conditions, pain, or seeking prevention of future injury. There are no child participants, as they are not candidates for the type of programs under investigation.

All data relating to the patient's physical therapy, diagnosis, co-morbidies, medical history, medications etc., will be used for analysis.

STUDY METHODS:

1. Describe how the data will be identified:

   Approved SpineZone staff will extract relevant outcomes data from the Electronic Medical Records system housed on a secure server. Identifiers will be stripped from the data, and claims will be indexed using Coding processes. Investigators will not have access to the pre-coded identifiers. Age, but not date of birth will be used, but no patients over the age of 89 will be included, thus it will not be an identifier. All systems used to store and view the data will be secure, with password protections and login access required. Once initial data extraction and de-identification is complete, the de-identified data will be stored on secure servers in a HIPAA compliant environment, and only transferred for biostatistics analytics through encrypted and password protected email to approved individuals (i.e. research biostatisticians) following a data use agreement.
2. Data that will be used:

Outcome variables: Validated questionnaire-based outcomes including but not limited to: VAS (visual analogue scale), ODI (oswestry disability index) for Low Back Pain, NDI (neck disability index) for neck pain, PSFS (patient specific functional scale), SBST (STarT Back Screening Tool), Hospital Anxiety and Depression Scale (HADS), medication usage (type, frequency), number of visits, progression to surgery (yes, no), dropout rates and reasons, Online compliance matrix(including access to educational material, log in rates, and self-reporting of compliance with workout regimen); physical examination measurements: strength and ROM measurements, and cost (based on procedural codes).

Predictor variables: Demographic, medical history, and treatment-specific variables including but not limited to: age, gender, ethnicity, diagnosis code (ICD-9/10), SpineZone rehabilitation diagnosis, treatment type, treatment history, radiologic diagnosis, duration of symptoms, postural factors, questionnaire-based pre-treatment disability, psychosocial status, prior treatments, concurrent treatments (e.g., nutrition, mindfulness), and pain scores.

d) Who will identify data to be reviewed:

SpineZone clinical staff and Principal Investigator

CONFIDENTIALITY OF DATA:

Data that is identified by the primary investigator for review will be additionally checked for any identifiers and stripped prior to analysis by biostatisticians. This data will be stored in two places. Initially, the de-identified data will be stored in the biostatistician's system for analysis. Once initial analysis is complete, the data will be loaded into a secure server with physical 24-hour security preventing unauthorized access to the hardware, with access to data only allowed through HTTPS login or through a direct and secure tunnel. Only investigators will have access to the login information.

Within two months of completion of the study, biostatisticians copy of the data will be destroyed. The data will be maintained in the secure hosted environment indefinitely.

Data will be transmitted with either password protection or PGP encryption on biostatistician computers. These computers and associated hardware are maintained in a secured facility with no public access. Computers are password protected and after 30 minutes of inactivity require the user to login again. Data and programs are backed up on a daily basis during the active phase of any project. Internet access is firewall protected. Anti-virus software is maintained (McAfee) with all incoming and outgoing documents scanned for viruses. Additionally, a scan of all files is performed daily.

Data storage will be on secure servers at a 24-hour guard facility, on windows server systems with updated enterprise virus protection software from Symantec. The database will only be accessible through an HTTPS log-in, with user-based access levels that ensure only personnel authorized by the principal investigator can gain access to the system. Any access will be tracked through a log of historical events that will track what user viewed or manipulated what data at any time.

Systems, security policies, and access logs will all be available for audit and review by the Principal Investigator at any time.

CONSENT:

Consent will be obtained in clinic, or through a form on an online portal for patients participating in the online treatment arm.

RISKS AND BENEFITS:

Risks: A confidentiality breach is a risk associated with data review research, however every measure will be instituted to ensure that patient information is kept confidential. Data analysis worksheets will be kept separate from EMR records. No subject PHI will be collected or shared.

Benefits: The participants are not likely to receive any benefit from the proposed research; however, society and investigators will benefit from the knowledge gained.

STATISTICAL CONSIDERATIONS:

As this is intended to be a data registry, no current statistical analyses are being proposed. Independent sub-studies utilizing data from this registry will be required to provide power analyses and proposed sample sizes necessary to carry out the objectives of the individual research question.

Data will be analyzed for individual sub-studies by biostatisticians located at the University of California, San Diego. All individuals participating in data analysis will be trained in research compliance, ethics, and will follow regulations according to the approved data use agreements in place.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* under 89 years of age
* Patients who have been prescribed physical rehabilitation for management of spine pain

Exclusion Criteria:

* under 18 years of age
* over 89 years of age
* Patients who are unable or medically unsafe to participate in physical rehabilitation for management of spine pain as determined by the prescribing physician

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Individuals between the ages of 18-89 who are seeking, or have been prescribed physical rehabilitation as a conservative management strategy for a complaint of spine pain (including, but not limited to neck pain, low back pain, thoracic spine pain, or scoliosis).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in pain: Visual Analogue Scale (VAS), 0-100mm | 3 months, 6 months, 1 year, and 2 years
  difference in VAS (in mm) between initial evaluation and endpoint
Change in disability (%) | 3 months, 6 months, 1 year, and 2 years
  difference in Neck Disability Index (for neck pain participants) or Oswestry Disability Index (for Low Back Pain participants), or Scoliosis Research Society Outcomes questionnaire-22 (for Scoliosis participants) between initial evaluation and endpoint
Change in quality of life | 3 months, 6 months, 1 year, and 2 years
  difference in EQ5-D (points) score between initial evaluation and endpoint
Change in strength (lbs*deg) | 3 months, 6 months, 1 year, and 2 years
  difference in spine extension torque as measured by isokinetic dynamometer between initial evaluation and endpoint
Change in Range of Motion (deg) | 3 months, 6 months, 1 year, and 2 years
  difference in total spine flexion and extension (in degrees) between initial evaluation and endpoint

SECONDARY OUTCOMES:
Change in spine extensor muscle cross sectional area (cm2) | 3 months
  Difference in cross sectional area of the multifidus and erector spinae muscles as measured via MRI between initial evaluation and endpoint
change in spine extensor muscle fatty infiltration (%) | 3 months
  difference in percentage of fat within the multifidus and erector spinae muscles as measured by T1-weighted MRI between initial evaluation and endpoint

OTHER OUTCOMES:
Change in medication usage (category) | 3 months, 6 months, 1 year, and 2 years
  difference in frequency of analgesic medication usage between initial evaluation and endpoint: frequency will be aggregated according to the following categories: [None, <1/day, 1-2/day, 3+/day]
Surgery (%) | 6 months, 1 year, and 2 years
  Percentage of participants that cross over into a surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Shahidi, P.T., Ph.D., Study Director — University of California, San Diego
Locations (1):
- SpineZone, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Patient data will only be accessible to SpineZone and collaborating research partners (UCSD)

REFERENCES:
- [Derived] Raiszadeh K, Tapicer J, Taitano L, Wu J, Shahidi B. In-Clinic Versus Web-Based Multidisciplinary Exercise-Based Rehabilitation for Treatment of Low Back Pain: Prospective Clinical Trial in an Integrated Practice Unit Model. J Med Internet Res. 2021 Mar 18;23(3):e22548. doi: 10.2196/22548. PMID 33734088